CLINICAL TRIAL: NCT01529424
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Response, Phase 2 Study of ISIS 304801 Administered Subcutaneously to Patients With Severe or Uncontrolled Hypertriglyceridemia
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of ISIS ApoC-III Rx in Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 304801-CS2
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Non-extensive PK/non post-prandial
  Interventions: Drug: ISIS apoC-III Rx; Drug: Placebo
- Group 2a (Experimental): Extensive PK
  Interventions: Drug: ISIS apoC-III Rx; Drug: Placebo
- Group 2b (Experimental): Post-prandial assessment
  Interventions: Drug: ISIS apoC-III Rx; Drug: Placebo
- Group 3 (Experimental): Stable dose of fibrate
  Interventions: Drug: ISIS apoC-III Rx; Drug: Placebo
- Group 4 (Experimental): Fredrickson Type 1 dyslipidemia
  Interventions: Drug: ISIS apoC-III Rx

INTERVENTIONS:
Drug: ISIS apoC-III Rx — Dose 1
  Arms: Group 1; Group 2a
Drug: ISIS apoC-III Rx — Dose 2
  Arms: Group 1; Group 2a; Group 2b; Group 3
Drug: ISIS apoC-III Rx — Dose 3
Drug: Placebo — Dose 1
  Arms: Group 1; Group 2a
Drug: Placebo — Dose 2
  Arms: Group 1; Group 2a; Group 2b; Group 3
Drug: Placebo — Dose 3
  Arms: Group 1; Group 2a; Group 2b; Group 3

SUMMARY:
The purpose of this study is to evaluate the dose/response pharmacodynamic effects of ISIS ApoC-III Rx vs. Placebo on fasting total apoC-III levels.

ELIGIBILITY:
Inclusion Criteria:

* Severe hypertriglyceridemia

Exclusion Criteria:

* HbA1c >/=9.0%, type 1 diabetes, or history of outpatient insulin use for more than 2 weeks in the last year
* Body mass index (BMI) >40 kg/m2
* History of bariatric surgery or currently on weight loss drugs
* Use of oral contraceptives or hormone replacement therapy or statins unless stable for 3 months prior to dosing
* Group 1 and 2 patients: Use of systemic corticosteroids, fibrates, niacin, fish oil or other products containing omega-3 fatty acids within 6 weeks of dosing. Group 3 patients: unable to discontinue use of systemic corticosteroids at least 6 weeks prior to dosing ; use of niacin, fish oil, or other products containing omega-3 fatty acids unless on a stable well controlled dose for at least 30 days prior to screening that is not anticipated to change during the study period. Group 4 patients: unable to discontinue use of systemic corticosteroids at least 6 weeks prior to dosing; use of fibrates niacin, fish oil, or other products containing omega-3 fatty acids unless on a stable well controlled dose for at least 30 days prior to screening that is not anticipated to change during the study period.
* Use of topical corticosteroids, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects unless dose is stable and well controlled for 30 days prior to dosing
* Any Screening laboratory values that are out of allowed reference ranges
* Inability to comply with protocol or study procedures
* Any other significant illness or condition that may adversely affect the subjects participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
VLDL apoC-III | 92 Days
  The effect of treatment with ISIS ApoC-III Rx or Placebo on fasting total apoC-III levels.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Farmville Internal Medicine, Farmville, North Carolina
  - Mark R. Cervi, Greenville, North Carolina
  - Physicians East, Quadrangle Medical Specialists, Greenville, North Carolina
  - Carolina East Family Medicine, Greenville, North Carolina
  - Eastern Carolina Physicians, Kinston, North Carolina
  - Natalie A Doyle, MD PA, Wilson, North Carolina
- Isis Investigational site, Chicoutimi, Quebec, Canada

REFERENCES:
- [Derived] Gaudet D, Alexander VJ, Baker BF, Brisson D, Tremblay K, Singleton W, Geary RS, Hughes SG, Viney NJ, Graham MJ, Crooke RM, Witztum JL, Brunzell JD, Kastelein JJ. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med. 2015 Jul 30;373(5):438-47. doi: 10.1056/NEJMoa1400283. PMID 26222559